CLINICAL TRIAL: NCT01956604
Title: The Oslo Study of Clonidine in Elderly Patients With Delirium
Acronym: LUCID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The inclusion rate was too low, due to the exclusion criteria.
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Bjørn Erik Neerland, MD, Medical doctor, PhD student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013-000815-26; 2013-000815-26 (EudraCT Number)
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clonidine (Experimental): Clonidine administered orally:
  Day 1/loading doses: 75µg every 3rd hour until maximum 4 doses. Day 2-7/maintenance doses: 75µg BID. Duration of treatment is maximum 7 days.
  Interventions: Drug: Clonidine
- Placebo (sugar pill) (Placebo Comparator): Placebo administered orally (identical capsula as for expirimental drug):
  Day 1/loading doases: 75µg every 3rd hour until maximum 4 doses. Day 2-7/maintenance doses: 75µg BID. Duration of treatment is maximum 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine
  Arms: Clonidine
Drug: Placebo
  Arms: Placebo (sugar pill)

SUMMARY:
Delirium ("acute confusional state")is characterized by an acute decline in attention and cognition, and is a common clinical syndrome in elderly patients.

The purpose of this randomised, controlled, parallel group pilot trial is to explore superiority of clonidine vs placebo in decreasing delirium in patients diagnosed delirium at the acute geriatric ward.

We will also study the feasibility of oral clonidine in a geriatric ward and effects of clonidine upon a variety of outcomes as a means to design a more definite study later.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 65 years old admitted to the Medical department
* Delirium or subsyndromal delirium diagnosed within the last 48 hours
* Signed informed consent from patient or relatives
* Expected cooperation of the patients for the treatment and follow up

Exclusion Criteria:

* Symptomatic bradycardia, bradycardia due to sick-sinus-syndrome, second- or third- degree AV-block (not treated With pacemaker) or any other reason causing HR <50 bpm at time of inclusion
* Symptomatic hypotension or orthostatic hypotension, or a systolic BP <120 at the time of inclusion
* Ischemic stroke within the last 3 months or critical peripheral ischemia
* Acute coronary syndrome, unstable or severe coronary heart disease (symptoms at minimal physical activity; NYHA 3 and 4) and moderate to severe heart failure (NYHA 3 and 4).
* A diagnosis of polyneuropathy or pheochromocytoma
* Renal insufficiency (estimated GFR<30 ml/min according to the MDRD formula).
* Body weight < 45 kg.
* Considered as moribund on admission.
* Not able to take oral medications
* Current use of tricyclic antidepressants, monoamine reuptake inhibitors or ciclosporin
* Previously included in this study
* Adverse reactions to clonidine or excipients (lactose, saccharose)
* Not speaking or reading Norwegian
* Any other condition as evaluated by the treating physician
* Admitted to the ICU

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
MDAS (Memorial delirium assessment scale) | Participants will be followed for the duration of hospital stay, an expected average of approximately 2 weeks

SECONDARY OUTCOMES:
Time-to-first delirium | 2 weeks
  We will compare the actively treated group with the placebo group (also with subanalyses for subsyndromal delirium and hypoactive/ hyperactive/ mixed delirium) with respect to:
  • time to first resolution, monitored by DSM-5 criteria
Incidence of "full-scale" delirium | 2 weeks
  • monitored by DSM-5 criteria
Severity of delirium | 2 weeks
  measured by MDAS, OSLA
Delirium subtype | 2 weeks
  Measured by MDAS, OSLA
The use of "rescue medication" | 2 weeks
Length of hospital stay | Hospital stay
Patient distress | 2 weeks
Side effects of clonidine | 4 months
Pharmacokinetic response to clonidine | 1 week
Pharmacodynamic response to clonidine | 2 weeks
Biomarkers | 2 weeks
Institutionalization | 4 months
Survival | 4 months
Cognitive function/ independence | 4 months

OTHER OUTCOMES:
Exposure-response analyses | 4 months
  We will also do per protocol analyses and exposure-response analyses based on measurements of the plasma concentration of clonidine

CONTACTS AND LOCATIONS:
Overall Officials: Torgeir Bruun Wyller, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Hov KR, Neerland BE, Andersen AM, Undseth O, Wyller VB, MacLullich AMJ, Skovlund E, Qvigstad E, Wyller TB. The use of clonidine in elderly patients with delirium; pharmacokinetics and hemodynamic responses. BMC Pharmacol Toxicol. 2018 Jun 8;19(1):29. doi: 10.1186/s40360-018-0218-1. PMID 29884231
- [Derived] Neerland BE, Hov KR, Bruun Wyller V, Qvigstad E, Skovlund E, MacLullich AM, Bruun Wyller T. The protocol of the Oslo Study of Clonidine in Elderly Patients with Delirium; LUCID: a randomised placebo-controlled trial. BMC Geriatr. 2015 Feb 10;15:7. doi: 10.1186/s12877-015-0006-3. PMID 25887557